CLINICAL TRIAL: NCT01400711
Title: Enhanced Recovery After Surgery (ERAS) Versus Conventional Postoperative Care in Patients Undergoing Major Intra-abdominal Surgery.
Brief Title: Enhanced Recovery After Surgery in Major Intrabdominal Procedures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Andrew's General Hospital, Patras, Greece (Other)
Responsible Party: Vassilios Alivizatos MD, Ph.D, St. Andrew General Hospital, Department of Surgery, Patra, Greece
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1VA
Record Dates: First submitted 2011-06-20; First posted 2011-07-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2010-08

CONDITIONS: Complication of Surgical and Medical Care.
Keywords: Fast-tract surgery, Enhanced recovery after surgery, multimodal surgery.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ERAS patients (Active Comparator): Patients planned to undergoing major intrabdominal surgery, following the ERAS perioperative care.
  Interventions: Other: ERAS perioperative care
- Control patients (Active Comparator): Patients planned to undergo major intrabdominal surgery, following the conventional perioperative care.
  Interventions: Other: Traditional

INTERVENTIONS:
Other: ERAS perioperative care — Patient's education before surgery, early mobilization and oral feeding after surgery, no opioids analgesics.
  Arms: ERAS patients
Other: Traditional — Nasogastric tube until bowel function, late oral eating, opioid analgesics.
  Arms: Control patients

SUMMARY:
Enhanced Recovery After Surgery (ERAS) programs have been introduced with aims of attenuating the stress response to surgery and enabling rapid recovery. There is strong evidence of the usefulness of the ERAS programs in patients undergoing colorectal surgery in terms of significantly reduced postoperative complications and shorter length of hospital stay, compared to the patients of traditional treatment. However, few studies exist about the implication of ERAS programs in major upper abdominal surgery patients.

The aim of this study was to compare morbidity, mortality and length of stay in patients undergoing major intrabdominal surgery, including upper and lower gastrointestinal, receiving either conventional postoperative care or an ERAS program.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* ASA grade < 4

Exclusion Criteria:

* Emergency surgery
* ASA grade > 3

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Morbidity. | 30 days after surgery

SECONDARY OUTCOMES:
Mortality. | 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- St. Andrew General Hospital, Department of Surgery, Pátrai, Greece

REFERENCES:
- [Result] Lassen K, Soop M, Nygren J, Cox PB, Hendry PO, Spies C, von Meyenfeldt MF, Fearon KC, Revhaug A, Norderval S, Ljungqvist O, Lobo DN, Dejong CH; Enhanced Recovery After Surgery (ERAS) Group. Consensus review of optimal perioperative care in colorectal surgery: Enhanced Recovery After Surgery (ERAS) Group recommendations. Arch Surg. 2009 Oct;144(10):961-9. doi: 10.1001/archsurg.2009.170. PMID 19841366